CLINICAL TRIAL: NCT05571657
Title: Understanding and Addressing the Disparity in Vaccination Coverage Among U.S. Adolescents Living in Rural Versus Urban Areas
Brief Title: COVID-19 Booster Dose Reminder/Recall for Adolescents
Acronym: AIMED COVID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Marshfield Clinic Research Foundation (Other)
Responsible Party: Principal Investigator, Huong McLean, PhD, Research Scientist, Marshfield Clinic Research Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MCL10517a; U01IP001093 (NIH)
Record Dates: First submitted 2022-10-06; First posted 2022-10-07 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: COVID-19 Vaccines
Keywords: reminder/recall; COVID-19; intervention; adolescents
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Reminder/recall
  Interventions: Behavioral: Reminder/Recall Sent Via Preferred Method of Communication
- Usual Care (No Intervention): No Reminder/Recall

INTERVENTIONS:
Behavioral: Reminder/Recall Sent Via Preferred Method of Communication — Parents of 12-17 year-old patients due for COVID-19 booster dose will receive a one-time vaccine reminder/recall via the parent's preferred method of communication (mailed letter, text message, email)
  Arms: Intervention

SUMMARY:
A single COVID-19 booster dose has been recommended in the United States for adolescents aged ≥12 years to enhance protection against SARS-CoV-2 infection. This study will assess the efficacy of a one-time reminder/recall for COVID-19 booster dose among eligible adolescents in a regional healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* Marshfield Clinic Health System patient aged 12-17 years with at least one preventive visit or two evaluation & management visits with a Marshfield Clinic Health System provider in the last 36 months
* Due for a COVID-19 booster dose (completed the COVID-19 primary series and it has been ≥5 months since their second dose)

Exclusion Criteria:

* Primary care provider is not affiliated with Marshfield Clinic Health System
* Opted out of Marshfield Clinic Health System centralized vaccine reminder notifications
* Received COVID-19 vaccine off label
* Missing or invalid contact information
* Deceased

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4304 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
COVID-19 Booster Dose | 90 days
  Number of patients that received a COVID-19 booster dose during follow-up based on electronic health data. Receipt of a COVID-19 booster dose within 90 days of randomization (yes/no) will be assessed using vaccination data available from the Marshfield Clinic Health System (MCHS) electronic health record, which includes vaccinations administered outside of MCHS through data exchanges with the Wisconsin Immunization Registry. Specifically patients will be classified as having received a COVID-19 booster dose if they have record of receipt of COVID-19 booster dose with a vaccination date during the 90-day follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Huong McLean, PhD, Principal Investigator — Marshfield Clinic Research Institute
Locations (1):
- Marshfield Clinic Health System, Marshfield, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/57/NCT05571657/Prot_000.pdf